CLINICAL TRIAL: NCT04066036
Title: Population Effectiveness of Dolutegravir Implementation in Sub-Saharan Africa: A Prospective Observational Cohort Study
Brief Title: Population Effectiveness of Dolutegravir Implementation in Sub-Saharan Africa
Acronym: DISCO
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Africa Health Research Institute (Other); Mbarara University of Science and Technology (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Wellcome Trust (Other); ViiV Healthcare (Industry); Harvard Medical School (HMS and HSDM) (Other); University of KwaZulu (Other); Emory University (Other)
Responsible Party: Principal Investigator, Mark Siedner, Associate Professor, Assistant Physician, Massachusetts General Hospital
Other Study IDs: 2019P000898-A; K23AI143470 (NIH); 212215 (Other Grant/Funding Number: ViiV Healthcare); WT108082AIA (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2019-08-21; First posted 2019-08-22 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: HIV-1-infection
Keywords: HIV Integrase Inhibitors; Sub-Saharan Africa; Anti-HIV Agents; Medication Adherence; Virologic Failure; Viral Drug Resistance; South Africa; Uganda; HIV-1
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, buffy coat, plasma, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: The study will enroll a total of 1,000 ART-experienced participants from the study sites in Uganda and South Africa who are being transitioned to TLD from non-nucleoside reverse transcriptase-based antiretroviral therapy.
  Interventions: Other: This is an observational study only.

INTERVENTIONS:
Other: This is an observational study only. — This is an observational study only.

SUMMARY:
This is a prospective observational cohort study enrolling participants in South Africa and Uganda who are prescribed an HIV treatment regimen containing lamivudine, tenofovir, and dolutegravir, which is known as TLD. We hope to better understand how effective TLD will be in sub-Saharan Africa. If treatment failure occurs, we seek to understand the possible reasons, including drug resistance and adherence challenges.

DETAILED DESCRIPTION:
This study is a prospective observational cohort study at three government-supported HIV clinics in rural South Africa and Uganda. We will enroll 1,000 adults living with HIV who are switched from first-line antiretroviral therapy (ART) containing non-nucleoside reverse transcriptase inhibitors (NNRTIs) to TLD. We will follow participants for one year with study visits at enrollment, 24 weeks, and 48 weeks. Study procedures include interviews, body measurements, chart review, and collection of blood and urine specimens for retrospective testing, including viral load, drug resistance testing, antiretroviral drug level testing, and tests to evaluate the effects of TLD on renal, liver, metabolic, and other organ function.

Aim 1: To determine the contributions of resistance prior to switch to TLD from a NNRTI-based regimen to risk of treatment failure after six and twelve months on TLD. Hypothesis: People living with HIV who experience virologic failure on TLD will have increased odds of NRTI mutations prior to TLD exposure, compared to controls with virologic suppression.

Aim 2: Explore pharmacologic measures of adherence to distinguish virologic failure on TLD due to suboptimal adherence versus resistance using 2a) urine tenofovir (TFV) levels and 2b) tenofovir diphosphate (TFV-DP) in dried blood spots (DBS). Hypothesis: Absence of TFV in urine and TFV-DP concentrations in DBS will distinguish ART failure with versus without resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* HIV-positive and in care at one of the study clinics
* Current use of NNRTI-based, first-line ART for a minimum of 6 months
* Prescribed change to TLD by clinic staff
* Residing within 100 kilometers of the treatment clinic without plans to change permanent residence in the next 48 weeks
* Consents to participation

Exclusion Criteria:

There are no specific exclusion criteria. Both men and women will be theoretically eligible. We note that decision to use TLD in patients at the recruitment clinic will be made by clinic staff, and referral for study procedures will not be made until after this decision is made. We also note that, as of the time of this protocol draft, TLD use might be limited to men, women of non-child bearing ages, and women confirmed to be on contraception. This study will follow both national guidelines and clinician discretion about use of TLD in the clinic population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll a total of 1,000 individuals from Uganda and South Africa, who are currently enrolled in care at one of the study clinics who have been taking NNRTI-based ART for a minimum of six months, and who are switching to TLD. 500 participants will be recruited from Uganda, and 500 will be recruited from South Africa.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with virologic failure (HIV-1 RNA >= 200 copies/mL) | 48 weeks
  HIV-1 RNA >= 200 copies/mL

SECONDARY OUTCOMES:
Proportion of participants with virologic failure (HIV-1 RNA >= 1,000 copies/mL) | 48 weeks
  HIV-1 RNA >= 1,000 copies/mL
Proportion of participants with HIV drug resistance | 24 and 48 weeks
  Proportion of participants with International AIDS Society-defined drug resistance mutations to their current regimen

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne M McCluskey, MD, Principal Investigator — Massachusetts General Hospital; Mark J Siedner, MD, MPH, Principal Investigator — Massachusetts General Hospital, Africa Health Research Institute
Locations (2):
- Africa Health Research Institute, Somkele, KwaZulu-Natal, South Africa
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Data will be made public and accessible through request after completion of the primary analysis.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After completion of the primary analysis
Access Criteria: De-identified data and supporting information will be made available upon request after agreement among the principal investigators, and based on what is allowable in the study informed consent documents.

REFERENCES:
- [Derived] McCluskey SM, Muyindike WR, Nanfuka V, Omoding D, Komukama N, Barigye IT, Kansiime L, Tumusiime J, Aung TN, Stuckwisch A, Hedt-Gauthier B, Marconi VC, Moosa MS, Pillay D, Giandhari J, Lessells R, Gupta RK, Siedner MJ. Population Effectiveness of Dolutegravir Implementation in Uganda: A Prospective Observational Cohort Study (DISCO), 48-Week Results. J Infect Dis. 2024 Sep 23;230(3):e622-e630. doi: 10.1093/infdis/jiae260. PMID 38748986